CLINICAL TRIAL: NCT02119819
Title: Comparison of the Oxyntomodulin Analog, LY2944876, to Once-Weekly Exenatide and to Placebo in Patients With Type 2 Diabetes
Brief Title: A Study to Compare a New Drug for Type 2 Diabetes to Placebo and to a Treatment Already Available for Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15062; 2013-003552-21 (EudraCT Number); I7I-MC-XNAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Weight loss
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Weight Loss | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 10 mg LY2944876 (Experimental): 10 milligrams (mg) LY2944876 given subcutaneously (SC) once weekly for 24 weeks.
  Participants remain on stable doses of metformin, as prescribed by their personal investigator if they were on metformin at study entry.
  Interventions: Drug: LY2944876; Drug: Metformin
- 15 mg LY2944876 (Experimental): 15 mg LY2944876 given SC once weekly for 24 weeks. Participants remain on stable doses of metformin, as prescribed by their personal investigator if they were on metformin at study entry.
  Interventions: Drug: LY2944876; Drug: Metformin
- 30 mg LY2944876 (Experimental): 30 mg LY2944876 given SC once weekly for 24 weeks. Participants remain on stable doses of metformin, as prescribed by their personal investigator if they were on metformin at study entry.
  Interventions: Drug: LY2944876; Drug: Metformin
- 50 mg LY2944876 (Experimental): 50 mg LY2944876 given SC once weekly for 24 weeks. Participants remain on stable doses of metformin, as prescribed by their personal investigator if they were on metformin at study entry.
  Interventions: Drug: LY2944876; Drug: Metformin
- Exenatide extended-release (Experimental): 2 mg exenatide extended-release given SC once weekly for 24 weeks. Participants remain on stable doses of metformin, as prescribed by their personal investigator if they were on metformin at study entry.
  Interventions: Drug: Exenatide extended-release; Drug: Metformin
- Placebo (Placebo Comparator): Placebo for LY2944876 and Exenatide given SC once weekly for 12 weeks. Participants assigned to placebo will have no injections during the second 12 weeks of the study.
  Participants remain on stable doses of metformin, as prescribed by their personal investigator if they were on metformin at study entry.
  Interventions: Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: LY2944876 — Administered SC
  Arms: 10 mg LY2944876; 15 mg LY2944876; 30 mg LY2944876; 50 mg LY2944876
Drug: Exenatide extended-release — Administered SC
  Arms: Exenatide extended-release
Drug: Placebo — Administered SC
  Arms: Placebo
Drug: Metformin — Oral

SUMMARY:
The main purpose of this study is to compare the safety and effectiveness of the study drug known as LY2944876 to exenatide extended-release and placebo in participants with type 2 diabetes mellitus. All drugs will be given by an injection under the skin. Participants remain on stable doses of metformin, as prescribed by their personal investigator if they were on metformin at study entry. Participants' involvement in the study is expected to last about 30 weeks.

DETAILED DESCRIPTION:
The study will include a 12 week blinded treatment period, where neither the participant nor the investigator will know to which treatment each individual is assigned. Thereafter follows a 12 week period where participants and the investigator will know which treatment they are assigned to. Participants' on LY2944876 and on exenatide extended-release continue treatment in this period, those who received placebo will be followed without treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with diabetes mellitus Type 2
* Have screening HbA1c ≥7.0% and ≤10.5% either on diet and exercise alone or on a stable dose of metformin (≥1000 mg/day) for 3 months prior to screening
* Have body mass index (BMI) ≥23 and ≤45 kilograms per meter squared at screening

Exclusion Criteria:

* Women of child bearing potential
* Participants who have used thiazolidinediones within 3 months prior to screening, or any other drugs for treatment of hyperglycemia (except metformin) within the prior 2 months
* Participants who have used insulin for diabetic control for more than 6 consecutive days within the prior year
* Participants with impaired renal function (serum creatinine >124 micromole per liter (µmol/L) [1.4 milligrams per deciliter (mg/dL)] in women, >133 µmol/L [1.5 mg/dL] in men)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (51):
- United States (31):
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Valley Endocrine, Fresno, Fresno, California
  - National Research Institute, Los Angeles, California
  - Desert Medical Group Inc, Palm Springs, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Encompass Clinical Research, Spring Valley, California
  - Meridien Research, Bradenton, Florida
  - M & O Clinical Research, LLC, Fort Lauderdale, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Compass Research, Oviedo, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - University of Hawaii, Honolulu, Hawaii
  - East West Medical Institute, Honolulu, Hawaii
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Iderc, P.L.C., Des Moines, Iowa
  - Cotton O'Neil Diabetes and Endocrinology Center, Topeka, Kansas
  - Mercy Medical Research Institute, Springfield, Missouri
  - St John's Mercy Medical Center, St Louis, Missouri
  - Mercy Health Research, Washington, Missouri
  - Southern New Hampshire Diabetes and Endocrinology, Nashua, New Hampshire
  - High Point Clinical Trials Center, High Point, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - The Corvallis Clinic P.C., Corvallis, Oregon
  - Blair Medical Associates, Inc., Altoona, Pennsylvania
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - San Gabriel Clinical Research, Georgetown, Texas
  - Oakwell Clinical Research, San Antonio, Texas
  - Southwest Health Associates, P.A., Sugar Land, Texas
  - Wade Family Medicine, Bountiful, Utah
- Greece (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ampelokipoi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampico
- Poland (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdynia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Puerto Rico (2):
  - Manati Medical Center, Manatí
  - American Telemedicine Center, San Juan
- Romania (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ploieşti
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timișoara

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 mg LY2944876: 10 milligrams (mg) LY2944876 given subcutaneously (SC) once weekly for 24 weeks, plus background PO metformin.
- 15 mg LY2944876: 15 mg LY2944876 given SC once weekly for 24 weeks, plus background PO metformin..
- 30 mg LY2944876: 30 mg LY2944876 given SC once weekly for 24 weeks, plus background PO metformin..
- 50 mg LY2944876: 50 mg LY2944876 given SC once weekly for 24 weeks, plus background PO metformin..
- Exenatide Extended-release: 2 mg exenatide extended-release given SC once weekly for 24 weeks, plus background PO metformin..
- Placebo: Placebo for LY2944876 and Exenatide given SC once weekly for 12 weeks,plus background PO metformin. Participants assigned to placebo will have no injections during the second 12 weeks of the study.
Period: Overall Study
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo
Started | 66 | 71 | 73 | 70 | 69 | 71
Completed | 57 | 66 | 69 | 63 | 62 | 56
Not Completed | 9 | 5 | 4 | 7 | 7 | 15
Not completed — Adverse Event | 3 | 1 | 2 | 3 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2 | 1 | 2
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 3 | 0 | 0 | 6 | 10
Not completed — Jury Duty | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Left the city to get a job | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 10 mg LY2944876: 10 milligrams (mg) LY2944876 given subcutaneously (SC) once weekly for 24 weeks.
- 15 mg LY2944876: 15 mg LY2944876 given SC once weekly for 24 weeks.
- 30 mg LY2944876: 30 mg LY2944876 given SC once weekly for 24 weeks.
- 50 mg LY2944876: 50 mg LY2944876 given SC once weekly for 24 weeks.
- Exenatide Extended-release: 2 mg exenatide extended-release given SC once weekly for 24 weeks.
- Placebo: Placebo for LY2944876 and Exenatide given SC once weekly for 12 weeks. Participants assigned to placebo will have no injections during the second 12 weeks of the study.
- Total: Total of all reporting groups
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo | Total
Number analyzed (Participants) | 66 | 71 | 73 | 70 | 69 | 71 | 420
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (9.4) | 59.0 (8.5) | 56.1 (8.3) | 55.6 (8.4) | 57.6 (9.1) | 56.5 (9.7) | 57.1 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 40 | 26 | 33 | 32 | 35 | 199
  Male | 33 | 31 | 47 | 37 | 37 | 36 | 221
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 21 | 26 | 19 | 22 | 22 | 129
  Not Hispanic or Latino | 42 | 42 | 42 | 47 | 44 | 47 | 264
  Unknown or Not Reported | 5 | 8 | 5 | 4 | 3 | 2 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 1 | 2 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 5 | 5 | 2 | 6 | 25
  White | 55 | 59 | 59 | 58 | 59 | 58 | 348
  More than one race | 6 | 6 | 8 | 6 | 6 | 6 | 38
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Greece | 6 | 6 | 5 | 4 | 5 | 6 | 32
  Puerto Rico | 1 | 2 | 2 | 1 | 3 | 3 | 12
  Romania | 9 | 10 | 10 | 9 | 9 | 10 | 57
  United States | 32 | 33 | 33 | 34 | 31 | 30 | 193
  Poland | 9 | 10 | 12 | 12 | 12 | 11 | 66
  Mexico | 9 | 10 | 11 | 10 | 9 | 11 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Week 12
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Baseline, Week 12
Population: All randomized participants with baseline and at least one post-baseline HbA1c data at Week 12. Missing observations are imputed using the Bayesian simple linear regression longitudinal model.
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo
Number analyzed (Participants) | 57 | 68 | 68 | 65 | 63 | 62
percentage of HbA1c | -1.07 (0.12) | -1.09 (0.11) | -1.44 (0.11) | -1.33 (0.11) | -1.42 (0.11) | -0.29 (0.11)
Statistical Analysis 1: Comparison: 10 mg LY2944876 vs Placebo; Test type: Superiority; p = 0.459, Bayesian; Posterior Mean Difference = -0.78, 90% CI 2-sided [-1.05 to -0.52], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: 15 mg LY2944876 vs Placebo; Test type: Superiority; p = 0.511, Bayesian; Posterior Mean Difference = -0.80, 90% CI 2-sided [-1.07 to -0.54], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: 30 mg LY2944876 vs Placebo; Test type: Superiority; p = 0.988, Bayesian; Posterior Mean Difference = -1.15, 90% CI 2-sided [-1.41 to -0.89], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: 50 mg LY2944876 vs Placebo; Test type: Superiority; p = 0.934, Bayesian; Posterior Mean Difference = -1.04, 90% CI 2-sided [-1.30 to -0.78], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: 10 mg LY2944876 vs Exenatide Extended-release; Test type: Superiority; p = 0.373, Bayesian; Posterior Mean Difference = 0.35, 90% CI 2-sided [0.08 to 0.61], Standard Error of Mean 0.16
Statistical Analysis 6: Comparison: 15 mg LY2944876 vs Exenatide Extended-release; Test type: Superiority; p = 0.433, Bayesian; Posterior Mean Difference = 0.33, 90% CI 2-sided [0.07 to 0.59], Standard Error of Mean 0.16
Statistical Analysis 7: Comparison: 30 mg LY2944876 vs Exenatide Extended-release; Test type: Superiority; p = 0.978, Bayesian; Posterior Mean Difference = -0.02, 90% CI 2-sided [-0.28 to 0.24], Standard Error of Mean 0.16
Statistical Analysis 8: Comparison: 50 mg LY2944876 vs Exenatide Extended-release; Test type: Superiority; p = 0.904, Bayesian; Posterior Mean Difference = 0.09, 90% CI 2-sided [-0.17 to 0.35], Standard Error of Mean 0.16

2. Secondary Outcome: Change From Baseline in HbA1c at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: All randomized participants with baseline and at least one post-baseline HbA1c data at Week 24. Missing observations are imputed using the Bayesian simple linear regression longitudinal model.
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo
Number analyzed (Participants) | 55 | 66 | 68 | 62 | 60 | 51
percentage of HbA1c | -0.85 (0.14) | -1.14 (0.13) | -1.37 (0.13) | -1.29 (0.13) | -1.48 (0.13) | -0.38 (0.14)

3. Secondary Outcome: Percent Change From Baseline in Body Weight
Time Frame: Baseline, Week 12; Baseline, Week 24
Population: All randomized participants with baseline and at least one post-baseline data for body weight. Missing observations are imputed using the Bayesian simple linear regression longitudinal model.
Measure: Mean (Standard Error); unit: Percentage change
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo
Number analyzed (Participants) | 57 | 68 | 68 | 65 | 63 | 63
Percentage change
  Week 12: number analyzed (Participants) | 57 | 68 | 67 | 65 | 63 | 63
  Week 12 | -1.09 (0.35) | -1.86 (0.33) | -2.01 (0.33) | -3.23 (0.34) | -2.04 (0.35) | -1.22 (0.34)
  Week 24: number analyzed (Participants) | 55 | 67 | 68 | 62 | 60 | 51
  Week 24 | -1.57 (0.47) | -2.13 (0.45) | -1.98 (0.45) | -3.41 (0.46) | -2.18 (0.47) | -1.70 (0.46)

4. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: Least square means (LSM) was calculated from mixed-effects model with repeated measures (MMRM) analysis using restricted maximum likelihood (REML) with metformin use, baseline body mass index (BMI) category, baseline HbA1c category, country, treatment, visit, and treatment-by-visit interaction as fixed effects, baseline fasting blood glucose as a covariate, and participant as a random effect.
Time Frame: Baseline, Week 12; Baseline, Week 24
Population: All randomized participants with baseline and at least one post-baseline data for fasting blood glucose. Missing observations are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo
Number analyzed (Participants) | 66 | 71 | 73 | 69 | 69 | 71
milligrams per deciliter (mg/dL)
  Week 12 | -20.881 (4.618) | -21.991 (4.371) | -31.309 (4.305) | -28.405 (4.506) | -39.074 (4.419) | -1.588 (4.519)
  Week 24 | -21.497 (4.919) | -30.186 (4.639) | -29.875 (4.548) | -31.390 (4.785) | -40.328 (4.726) | 0.124 (4.973)

5. Secondary Outcome: Change From Baseline in 7-point Self-Monitored Blood Glucose (SMBG) Values
Description: SMBG 7-point profiles were measured at morning pre-meal, morning 2 hours post-meal, mid-day pre-meal, mid-day 2 hours post-meal, evening pre-meal, evening 2 hours post-meal, and at bedtime. LSM were calculated from MMRM analysis using REML with metformin use, baseline BMI category, baseline HbA1c category, country, treatment, visit, and treatment-by-visit interaction as fixed effects, baseline fasting blood glucose as a covariate, and participant as a random effect.
Time Frame: Baseline, Week (Wk) 12; Baseline, Week 24
Population: All randomized participants with baseline and at least one post-baseline data for SMBG. Missing observations are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo
Number analyzed (Participants) | 66 | 71 | 73 | 69 | 69 | 71
mg/dL
  Morning pre-meal (Week 12) | -26.8 (3.9) | -28.4 (3.8) | -34.3 (3.7) | -34.8 (3.8) | -38.7 (3.8) | -7.4 (3.8)
  Morning pre-meal (Week 24) | -23.5 (4.7) | -29.1 (4.5) | -29.6 (4.3) | -34.2 (4.5) | -36.8 (4.5) | -14.4 (4.9)
  Morning 2 hours post-meal (Week 12) | -27.9 (6.7) | -34.2 (6.8) | -36.0 (6.3) | -26.4 (6.6) | -43.5 (6.5) | -1.5 (6.5)
  Morning 2 hours post-meal (Week 24) | -29.9 (6.5) | -35.9 (6.5) | -37.1 (6.1) | -42.8 (6.4) | -42.7 (6.4) | -6.3 (6.8)
  Mid-day pre-meal (Week 12) | -17.1 (5.1) | -19.6 (5.1) | -26.1 (4.8) | -24.2 (5.0) | -23.5 (5.0) | -2.3 (5.0)
  Mid-day pre-meal (Week 24) | -16.3 (5.6) | -23.4 (5.6) | -22.4 (5.3) | -23.5 (5.4) | -23.9 (5.5) | -4.0 (6.0)
  Mid-day 2 hours post-meal (Week 12) | -17.1 (6.4) | -20.7 (6.3) | -24.6 (6.0) | -22.2 (6.2) | -27.4 (6.2) | -8.9 (6.1)
  Mid-day 2 hours post-meal (Week 24) | -12.2 (6.1) | -26.6 (5.9) | -21.9 (5.7) | -33.4 (5.9) | -37.2 (5.9) | -8.5 (6.4)
  Evening pre-meal (Week 12) | -24.1 (5.3) | -24.8 (5.2) | -28.5 (4.9) | -30.1 (5.1) | -24.7 (5.1) | -1.5 (5.1)
  Evening pre-meal (Week 24) | -24.9 (5.7) | -24.3 (5.6) | -33.0 (5.3) | -29.6 (5.4) | -36.4 (5.6) | -5.7 (6.0)
  Evening 2 hours post-meal (Week 12) | -25.1 (5.9) | -26.5 (5.7) | -33.4 (5.4) | -32.8 (5.7) | -33.5 (5.7) | 4.0 (5.6)
  Evening 2 hours post-meal (Week 24) | -30.2 (5.9) | -27.9 (5.8) | -26.0 (5.5) | -37.2 (5.8) | -36.9 (5.8) | 1.1 (6.2)
  Bedtime (Week 12) | -19.3 (5.7) | -33.5 (5.8) | -33.2 (5.8) | -36.2 (5.6) | -41.6 (5.7) | 5.6 (5.7)
  Bedtime (Week 24) | -28.9 (6.0) | -25.4 (6.0) | -32.3 (5.7) | -38.5 (5.9) | -42.9 (6.0) | -6.9 (6.4)

6. Secondary Outcome: Change From Baseline in Lipids
Description: Change from baseline in high-density lipoprotein cholesterol (HDL-C), total cholesterol, triglycerides, and low-density lipoprotein cholesterol (LDL-C). LSM was calculated from MMRM analysis using REML with metformin use, baseline BMI category, baseline HbA1c category, country, treatment, visit, and treatment-by-visit interaction as fixed effects, baseline parameter result as a covariate, and participant an a random effect.
Time Frame: Baseline, Week 24
Population: All randomized participants with baseline and at least one post-baseline data for lipids. Missing observations are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo
Number analyzed (Participants) | 66 | 71 | 73 | 69 | 69 | 71
mg/dL
  HDL-C | 1.56 (1.03) | 0.92 (0.98) | 0.90 (0.96) | 1.04 (1.01) | 2.35 (0.990) | 2.17 (1.04)
  Total Cholesterol | -1.26 (4.37) | -1.12 (4.16) | -1.46 (4.09) | -5.11 (4.24) | -0.12 (4.22) | 7.32 (4.40)
  Triglycerides | -14.63 (11.49) | -13.32 (10.93) | -15.40 (10.59) | -20.96 (11.16) | -11.83 (11.01) | 10.61 (11.58)
  LDL-C | -1.37 (3.75) | -0.40 (3.57) | -0.24 (3.56) | -0.04 (3.72) | 0.37 (3.65) | 4.55 (3.81)

7. Secondary Outcome: Change From Baseline in Fasting Fibroblast Growth Factor 21
Description: LSM was calculated from MMRM analysis using REML with metformin use, baseline BMI category, baseline HbA1c category, country, treatment, visit, and treatment-by-visit interaction as fixed effects, baseline parameter result as a covariate, and participant as a random effect.
Time Frame: Baseline, Week 12; Baseline, Week 24
Population: All randomized participants with baseline and at least one post-baseline data for fasting fibroblast growth factor 21. Missing observations are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: microgram per liter (µg/L)
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo
Number analyzed (Participants) | 66 | 71 | 73 | 69 | 69 | 71
microgram per liter (µg/L)
  Week 12 | -0.07 (0.071) | 0.06 (0.068) | -0.03 (0.068) | -0.14 (0.069) | -0.09 (0.069) | -0.11 (0.071)
  Week 24 | 0.06 (0.071) | -0.04 (0.068) | -0.07 (0.067) | -0.12 (0.070) | -0.06 (0.069) | -0.09 (0.073)

8. Secondary Outcome: Percentage of Participants Requiring Rescue Therapy
Description: Participants who received rescue medication with non-study antihyperglycemic medications or change their stable dose of metformin.
Time Frame: Baseline through Therapy Completion (Week 24)
Population: All randomized participants with baseline and at least one post-baseline data for participants requiring rescue therapy.
Measure: Number; unit: percentage of participants
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo
Number analyzed (Participants) | 66 | 71 | 73 | 69 | 69 | 71
percentage of participants | 6.1 | 2.8 | 2.7 | 4.3 | 2.9 | 11.3

9. Secondary Outcome: Percentage of Participants Developing Anti-Drug Antibodies to LY2944876
Description: Percentage of participants developing anti-drug antibodies to LY2944876.
Time Frame: Week 12 and Week 24
Population: All randomized participants who received study drug and had evaluable immunogenicity.
Measure: Number; unit: percentage of participants
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo
Number analyzed (Participants) | 66 | 71 | 73 | 70 | 69 | 71
percentage of participants
  Week 12: number analyzed (Participants) | 58 | 69 | 68 | 65 | 64 | 64
  Week 12 | 1.7 | 1.4 | 1.5 | 0 | 1.6 | 0
  Week 24: number analyzed (Participants) | 57 | 67 | 68 | 60 | 63 | 57
  Week 24 | 1.8 | 0 | 1.5 | 0 | 0 | 0

10. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY2944876
Description: Evaluable pharmacokinetic concentrations from the specified timepoints were combined and utilized in a population approach to determine the population mean estimate and standard deviation at steady-state.
Time Frame: Baseline, Week 8, Week 12, Week 16, Week 20, Week 24
Population: All randomized participants who received study drug LY2944876 and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876
Number analyzed (Participants) | 66 | 71 | 73 | 70
nanogram per milliliter (ng/mL) | 607 (282) | 799 (368) | 1690 (732) | 2570 (1240)

11. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) of LY2944876
Description: as for outcome 10
Time Frame: Baseline, Week 8, Week 12, Week 16, Week 20, Week 24
Population: All randomized participants who received study drug LY2944876 and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876
Number analyzed (Participants) | 66 | 71 | 73 | 70
nanograms*hour per milliliter (ng*h/mL) | 88100 (40600) | 117000 (50800) | 247000 (106000) | 381000 (187000)

12. Secondary Outcome: Change From Baseline in Adiponectin Levels
Description: LSM are calculated from MMRM analysis using REML with metformin use, baseline BMI category, baseline HbA1c category, country, treatment, visit, and treatment-by-visit interaction as fixed effects, baseline parameter result as a covariate, and participant as a random effect.
Time Frame: Baseline, Week 12; Baseline, Week 24
Population: All randomized participants with baseline and at least one post-baseline data for adiponectin levels. Missing observations are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: µg/L
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo
Number analyzed (Participants) | 66 | 71 | 73 | 69 | 69 | 71
µg/L
  Week 12 | 0.14 (0.168) | 0.03 (0.160) | -0.10 (0.157) | 0.12 (0.161) | 0.04 (0.160) | 0.03 (0.164)
  Week 24 | 0.03 (0.245) | 0.30 (0.226) | 0.28 (0.221) | 0.58 (0.235) | 0.14 (0.231) | 0.25 (0.250)

13. Secondary Outcome: Change From Baseline in Beta-Hydroxy Butyrate Levels
Description: as for outcome 12
Time Frame: Baseline, Week 12; Baseline, Week 24
Population: All randomized participants with baseline and at least one post-baseline data for beta-hydroxy butyrate levels. Missing observations are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo
Number analyzed (Participants) | 66 | 71 | 73 | 69 | 69 | 71
mg/dL
  Week 12 | -0.27 (0.13) | -0.28 (0.12) | -0.13 (0.12) | -0.31 (0.12) | -0.29 (0.12) | -0.23 (0.13)
  Week 24 | -0.33 (0.11) | -0.39 (0.10) | -0.34 (0.10) | -0.33 (0.10) | -0.19 (0.10) | -0.37 (0.11)

14. Secondary Outcome: Change From Baseline in Glucagon Levels
Description: as for outcome 12
Time Frame: Baseline, Week 12; Baseline, Week 24
Population: All randomized participants with baseline and at least one post-baseline data for glucagon levels. Missing observations are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: picomol per liter (pmol/L)
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo
Number analyzed (Participants) | 66 | 71 | 73 | 69 | 69 | 71
picomol per liter (pmol/L)
  Week 12 | -1.26 (0.82) | -2.65 (0.79) | -5.14 (0.79) | -6.21 (0.81) | -1.58 (0.79) | -0.04 (0.84)
  Week 24 | -2.30 (1.15) | -2.25 (1.05) | -4.40 (1.05) | -4.93 (1.11) | -0.19 (1.08) | 0.66 (1.16)

15. Secondary Outcome: Change From Baseline in Insulin Levels
Description: as for outcome 12
Time Frame: Baseline, Week 12; Baseline, Week 24
Population: All randomized participants with baseline and at least one post-baseline data for insulin levels. Missing observations are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: micro-international units/milliliter
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo
Number analyzed (Participants) | 66 | 71 | 73 | 69 | 69 | 71
micro-international units/milliliter
  Week 12 | 0.30 (1.21) | 0.97 (1.13) | 0.03 (1.14) | 0.96 (1.17) | 2.78 (1.14) | -0.85 (1.16)
  Week 24 | -1.44 (1.51) | 0.68 (1.39) | 0.58 (1.40) | 0.34 (1.48) | 1.97 (1.40) | 1.45 (1.51)

ADVERSE EVENTS:
Description: All randomized participants who received at least 1 dose of study drug.
Arm/Group | 10 mg LY2944876 | 15 mg LY2944876 | 30 mg LY2944876 | 50 mg LY2944876 | Exenatide Extended-release | Placebo
Serious Adverse Events (participants affected / at risk) | 0/66 | 2/71 | 2/73 | 3/70 | 3/69 | 2/71
Other Adverse Events (participants affected / at risk) | 34/66 | 47/71 | 39/73 | 46/70 | 38/69 | 16/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg LY2944876 (N=66) | 15 mg LY2944876 (N=71) | 30 mg LY2944876 (N=73) | 50 mg LY2944876 (N=70) | Exenatide Extended-release (N=69) | Placebo (N=71)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Branchial cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel perforation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg LY2944876 (N=66) | 15 mg LY2944876 (N=71) | 30 mg LY2944876 (N=73) | 50 mg LY2944876 (N=70) | Exenatide Extended-release (N=69) | Placebo (N=71)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (7) | 3 (3) | 4 (5) | 1 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4) | 4 (4) | 5 (8) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (35) | 15 (24) | 13 (45) | 12 (25) | 18 (52) | 4 (16)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 5 (8) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (28) | 21 (33) | 20 (53) | 32 (90) | 17 (55) | 4 (4)
Vomiting (Gastrointestinal disorders) | 8 (9) | 6 (6) | 10 (21) | 22 (37) | 6 (12) | 2 (3)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 4 (5) | 1 (3) | 2 (2) | 1 (1) | 2 (3)
Nasopharyngitis (Infections and infestations) | 8 (8) | 9 (11) | 5 (5) | 4 (4) | 6 (7) | 2 (3)
Sinusitis (Infections and infestations) | 1 (1) | 5 (6) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 10 (12) | 5 (5) | 3 (3) | 4 (4) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (6) | 1 (2) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 4 (4) | 2 (2) | 2 (2) | 5 (9) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 6 (6) | 6 (6) | 8 (9) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (7) | 1 (1) | 2 (2) | 2 (3) | 2 (3)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 5 (7) | 9 (13) | 5 (5) | 6 (11) | 9 (14) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days